CLINICAL TRIAL: NCT06800001
Title: Efficacy of Physical Activity for the Management of Stereotyped Behavior and Anxiety in Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Efficacy of Physical Activity for the Management of Stereotyped Behavior and Anxiety in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Saba Rashid, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2024/97
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder (ASD); Stereotyped Behavior; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Stereotyped Behavior; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Who receives intervention i.e Physical Activity Intervention (Experimental)
  Interventions: Other: Physical Activity
- Who would receive intervention after study completion (Active Comparator)
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Physical Activity — Physical Activity is an 8-week practical intervention for managing the stereotyped behavior & anxiety. Week 1: Introduction - Build engagement with the help of rapport building. Learn & practice ball-tapping exercise with warm up & cool down relaxation exercise. Week 2: Calmness- Practice jumping in trampoline exercise and learn balloon breathing exercise that give calmness. Week 3: Focus enhancement-Learn skills of jumping exercise to increase focus and improve impulse. Week 4: Strength, balance, and stress relief -explore the gym ball exercise in different directions that improves emotional regulation. Week 5: self control - Learn strategies for specific jumping patterns that improves impulse control and focus in children with ASD. Week 6: Reduce Stereotyped Behaviors - Learn complex trampoline exercises. Week 7: Skill Reinforcement- Review exercises, increasing speed or direction changes. Week 8: Integration -Encourage playful interaction to maintain engagement & consolidate skills.

SUMMARY:
The primary purpose of the study is to investigate whether physical activity can significantly manage stereotyped behavior and anxiety in children diagnosed with Autism Spectrum Disorder (ASD). The study aims to contribute to the existing literature by providing robust evidence on the efficacy of Physical Activity intervention for ASD, which could inform clinical practices and improve treatment outcomes.

DETAILED DESCRIPTION:
The current quantitative study will be carried out in two phases. A cross-sectional survey will assess the autism category (mild, moderate and severe), stereotyped behavior and anxiety in autistic children during the first phase. A randomized controlled trial (RCT) will be done during the second phase where children with Autism Spectrum Disorder who are identified with moderate category of autism, stereotyped behavior and anxiety will be categorized into two groups i.e. waitlist control group and intervention group through the process of randomization. Then physical activity intervention would be applied to participants in the intervention group. The control group is the waitlist control group so initially no intervention will be given to participants in the control group but the intervention will be given to the control group participants once the study is completed. The physical activity intervention would be implemented on participants using individual and in-person modes. The pre-and post-assessment will be done at Times 1 and 2 within and between control and interventional groups. After doing post assessment the difference between pre and post-assessment will be compared to explore the efficacy of physical activity intervention in children with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

Autistic children who are students of special education school. Only autistic children age 8 to 12 are part of the study. The participants who completed the informed consent will be part of the study. Participants who were showing symptoms of mild to moderate level of autistic symptoms as assessed by childhood autism rating scale. Participants should not have any physical or other mental health condition that would Prevent them from engaging in physical activity sessions safely were part of this study.

Exclusion Criteria:

Adults students are not part of the study. Autistic children who are not part of special education school. The participants who are severe autism category not part of the study. The participants who are under serious clinical condition will not be part of study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale | 3 months
  CARS consists of 15 items that assess various aspects of a child's behavior, including social interaction, communication, repetitive behaviors on the autism spectrum. CARS scored on a scale of 15-60, with higher scores indicating more severe autism. The Scoring following:
  15-29.5: Non-autistic 30-36.5: Mild to moderate autism 37-60: Severe autism

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rashid, MPhil Scholar, Principal Investigator — Fatima Jinnah Women University, Rawalpindi, Pakistan
Locations (1):
- Vive Pricinipal ASEA, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical concerns the data will not be shared. All research findings will be published in aggregate form maintaining participants anonymity.

REFERENCES:
- [Background] Ferreira JP, Ghiarone T, Junior CRC, Furtado GE, Carvalho HM, Rodrigues AM, Toscano CVA. Effects of Physical Exercise on the Stereotyped Behavior of Children with Autism Spectrum Disorders. Medicina (Kaunas). 2019 Oct 14;55(10):685. doi: 10.3390/medicina55100685. PMID 31615098
- See also: Related Info — https://link.springer.com/article/10.1007/s40489-023-00418-x